CLINICAL TRIAL: NCT02912585
Title: Oropharyngeal Administration of Colostrum and Prevention of Infections in Very Low Birthweight Infants
Brief Title: Oropharyngeal Administration of Colostrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Daniela Marques de Lima Mota Ferreira, Principal Investigator / Professor of Pediatrics / Head of Neonatology Division, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CEP 333.886
Record Dates: First submitted 2016-07-27; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Health Behavior
Keywords: colostrum
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Own mother's colostrum (Experimental): Oropharyngeal administration of own mother's colostrum.
  Interventions: Biological: Oropharyngeal administration of own mother's colostrum
- Placebo (Placebo Comparator): Oropharyngeal administration of sterile water.
  Interventions: Other: Oropharyngeal administration of sterile water (placebo)
- Donor human milk (Active Comparator): Oropharyngeal administration of donor human milk.
  Interventions: Biological: Oropharyngeal administration of donor human milk

INTERVENTIONS:
Biological: Oropharyngeal administration of own mother's colostrum
  Other Names: OMC Group
  Arms: Own mother's colostrum
Other: Oropharyngeal administration of sterile water (placebo)
  Other Names: Placebo Group
  Arms: Placebo
Biological: Oropharyngeal administration of donor human milk
  Other Names: DHM Group
  Arms: Donor human milk

SUMMARY:
Infections are the main causes of morbidity and mortality in very low birth weight infants. Use of mother's own breast milk in feeding these babies is associated with a decreased risk of acquiring nosocomial infection. This protective effect is assigned to a plurality of immune components in human milk. However, clinical instability of the preterm newborn in the first days of life results in delayed initiation of enteral nutrition. Thus, alternative methods for colostrum administration have been investigated, such as oropharyngeal administration with evidence that would be safe and feasible to perform in children admitted to the NICU in the first hours of life. Objective: To evaluate the immune stimulatory effect of oropharyngeal administration of colostrum in the incidence of sepsis in very low birth weight preterm infants.

DETAILED DESCRIPTION:
Background: Infections are the main causes of morbidity and mortality in very low birth weight infants. Use of mother's own breast milk in feeding these babies is associated with a decreased risk of acquiring nosocomial infection. This protective effect is assigned to a plurality of immune components in human milk. However, clinical instability of the preterm newborn in the first days of life results in delayed initiation of enteral nutrition. Thus, alternative methods for colostrum administration have been investigated, such as oropharyngeal administration with evidence that would be safe and feasible to perform in children admitted to the NICU in the first hours of life.

Objective: To evaluate the immune stimulatory effect of oropharyngeal administration of colostrum in the incidence of sepsis in very low birth weight preterm infants.

Methods: This was a prospective, randomized and blind study that included infants less than 34 weeks gestational age and birth weight less than 1,500 g, from 15 July 2013 to 15 July 2015.

The babies were divided initially into two groups for oropharyngeal administration or not of mother's own milk: Group 1 - underwent oropharyngeal administration of mother's own milk of and Group 2 - underwent oropharyngeal administration of sterile water, considered an inert substance. Newborns who were drawn to the Group 1 and it was not possible to obtain sufficient mother's own milk volume constituted a third group called Group 3 that receive oropharyngeal administration of donor breast milk. Oropharyngeal administration were initiated within the first 48-72 hours of life and maintained for 48 hours. Before the oropharyngeal administration, 24 hours after and 14 days after, samples of blood and urine were collected from the newborns to IgA and lactoferrin dosage.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight < 1500 g and gestational age < 34 weeks

Exclusion Criteria:

* congenital anomalies
* gastrointestinal disorders
* maternal history of substance abuse or positive maternal HIV status.

Ages: 72 Hours to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2013-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of late-onset sepsis | an average of 3 months
  Number of participants with late-onset sepsis
Measurement of immunologic factors in urine and blood samples using enzyme-linked immunoassay (ELISA). | an average of 3 months
  ELISA Index of immunologic factors in urine and blood samples

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferreira DMLM, Oliveira AMM, de Leves DV, de Bem EB, Fatureto GG, Navarro NF, Afonso NG, Santiago FM, Mineo JR, Sopelete MC, Martinez FE, Bernardino Neto M, Abdallah VOS. Randomized Controlled Trial of Oropharyngeal Colostrum Administration in Very-low-birth-weight Preterm Infants. J Pediatr Gastroenterol Nutr. 2019 Jul;69(1):126-130. doi: 10.1097/MPG.0000000000002356. PMID 30964820